CLINICAL TRIAL: NCT03242486
Title: Safety and Effectiveness Evaluation of Toric Intraocular Lens
Brief Title: Clinical Evaluation of Toric Intraocular Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nidek Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TIOL-YST
Record Dates: First submitted 2017-06-16; First posted 2017-08-08 (Actual); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Cataract; Astigmatism
MeSH Terms: conditions — Cataract; Astigmatism

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- toric intraocular lens (Experimental): toric intraocular lens is implanted to all subjects
  Interventions: Device: toric intraocular lens

INTERVENTIONS:
Device: toric intraocular lens

SUMMARY:
Evaluate efficacy and safety of the toric IOL implanted into aphakic eye with corneal astigmatism after cataract surgery.

DETAILED DESCRIPTION:
Effectiveness

* primary endpoint is visual acuity with pre-determined spherical correction.
* secondary endpoint is UCVA with spherical correction, BSCVA, Refractive Cylinder Correction, Spherical Equivalent, IOL rotation

Safety

* number and percentage of adverse event

ELIGIBILITY:
Inclusion Criteria:

* Patients with age of 40 years or older
* Patients with age-related cataract in one eye or both eyes.
* Patients willing to participate in the required postoperative study.
* Patient who can understand and sign the consent document.
* An eye whose pupil diameter after mydriasis is 5 mm or greater.
* An eye whose preoperative corneal cylindrical power is 1.0D or more.
* An eye whose postoperative astigmatism is predicted to be less than 0.5 D.
* An eye whose postoperative visual acuity with spherical addition is 0.8 D or more.

Exclusion Criteria:

* Disorder of corneal endothelium
* Uncontrolled glaucoma
* Active Uveitis
* Diabetic retinopathy
* Retinal detachment
* Congenital ocular anomalies
* Choroidal hemorrhage
* Shallow anterior chamber
* Microphthalmus
* Corneal dystrophy
* Optic atrophy
* Ocular hypertension
* Amblyopia
* Previous history of corneal transplantation
* Active Iritis
* Corneal disorder
* Macular degeneration
* Retinal degeneration
* Clinically significant change in macula and/or retinal pigment epithelium
* Corneal irregular astigmatism
* Atopic disease
* Brittleness of Zinn's zonule, fractured zonule and lens luxation (including subluxation)
* Pseudo-exfoliation syndrome
* Iris neovascularization
* Long axis length eye (axis length : 28mm or more)
* Severe dry eye, abnormality of the lens surface
* Concurrent participation in another drug and device clinical investigation
* Patient with mental deficiency or psychiatric disorder and/or who is not capable of expressing the consent of participating in the trial
* Patient who is judged inappropriate by investigators or sub-investigators

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Visual acuity | postoperative 6 months
  Visual acuity with pre-determined spherical correction

SECONDARY OUTCOMES:
Visual acuity | postoperative 6 months
  UCVA with spherical correction, BSCVA, Refractive Cylinder Correction, Spherical Equivalent
IOL rotation | postoperative 6 months
  angle of rotation

OTHER OUTCOMES:
Adverse events | one year
  Severity and causal relationship

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sugita I, Ogawa T, Ichikawa K, Okita T, Negishi K, Nakano T, Tsuneoka H. Rotational stability and clinical outcomes of a new one piece toric intraocular lens with anchor-wing haptics. BMC Ophthalmol. 2022 Jan 15;22(1):26. doi: 10.1186/s12886-021-02240-7. PMID 35033047